CLINICAL TRIAL: NCT03365180
Title: Starter Kit Study in Insulin naïve Patients With Type 2 Diabetes
Brief Title: Starter Kit Study in Insulin naïve Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Signe Schmidt (Other)
Collaborators: Technical University of Denmark (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Signe Schmidt, Principal Investigator, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StarterKit2017
Record Dates: First submitted 2017-09-06; First posted 2017-12-07 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Starter Kit Algorithm (Experimental): Basal insulin initiation and titration using the Starter Kit Algorithm at two weeks, followed by standard of care titration during the following the next 10 weeks (maximum), or until optimal daily dose is considered identified.
  Interventions: Device: Starter Kit Algorithm

INTERVENTIONS:
Device: Starter Kit Algorithm — Long acting insulin titration to target

SUMMARY:
The concept consists of an initial period (two weeks) of intensive data capture by use of continuous glucose monitoring (CGM) during basal insulin initiation, followed by a second period (variable duration) of basal insulin titration guided by self monitored blood glucose. Data captured during the first period are used as input to an algorithm that estimates the optimal daily dose for the individual patient. The estimated optimal daily dose is used to guide the titration of the basal insulin during the second period. The goal is to safely and successfully achieve blood glucose targets. The concept is based on the use of basal insulin degludec (Tresiba, Novo Nordisk A/S).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 18-75 years
* HbA1c 53-86 mmol/mol (7.0-10.0%)
* BMI 20-40 kg/m2
* Insulin-naïve
* Willingness to use CGM consistently during the study period and send/receive data and dose advice to/from HCP via a mobile phone
* Signed informed consent prior to any study procedures

Exclusion Criteria:

* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Active proliferative retinopathy
* Mean blood glucose > 15 mmol/l the week prior to screening
* Blood glucose > 20 mmol/l on the screening day
* Non-fasting ketones > 0,5 mmol/l on the screening day
* Use of sulfonylurea within 14 days prior to or during the study period
* Change in other antidiabetic medicine than basal insulin during the study period
* Use of corticosteroids within 30 days prior to or during the study period
* Marked change in lifestyle within 30 days prior to or during the study period as assessed by the investigator
* People with type 2 diabetes that suffer from conditions which make tight diabetes control undesirable, e.g. severe cardiovascular disease, according to the investigator
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation
* Overall treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of estimate 1 | through study completion, 12 weeks
  Accuracy of the estimated optimal daily dose (calculated by the Starter Kit algorithm based on continuous glucose monitoring (CGM) data collected during day 1-14) compared with the observed optimal daily dose in percentage deviation.
  In this context, optimal daily dose is the dose considered to keep fasting glucose levels below 6 mmol/L.
Accuracy of estimate 2 | through study completion, 12 weeks
  The number of estimated optimal daily doses by the Starter Kit Algorithm at two weeks that fall within a patient specific confidence interval.
  The confidence interval is determined using the Starter Kit Algorithm at the end of study, one interval for each patient.
  Upper boundary: the optimal daily dose estimated to bring lowest hour of CGM values within a day to 4.0 mmol/L Lower boundary: the optimal daily dose estimated to bring lowest hour of CGM values within a day to 6.0 mmol/L

SECONDARY OUTCOMES:
Accuracy of estimate 3 | through study completion, 12 weeks
  Accuracy of the estimated optimal daily dose (calculated based on self-monitored blood glucose data collected during day 1-14) compared with the observed optimal daily dose.
Number of patients in glucose target | through study completion, 12 weeks
  Number of participants in target at end of study
Algorithm deviations | 12 weeks (total duration of study)
  Number of titration algorithm deviations due to risk of hypoglycemia (based on evaluation of CGM data)
Quality of treatment 1 | through study completion, 12 weeks
  Qualitative assessment by the investigator of participants who do not reach the observed optimal daily dose within 12 weeks: Frequency of participants who are in need of additional basal insulin to achieve the target blood glucose.
Quality of treatment 2 | through study completion, 12 weeks
  Qualitative assessment by the investigator of participants who do not reach the observed optimal daily dose within 12 weeks: Frequency of participants who are in need of additional drugs to achieve the target blood glucose.
Number of self-monitored blood glucose values ≤3.9 mmol/L | 12 weeks (total duration of study)
  Number of self-monitored blood glucose values ≤3.9 mmol/L
Number of self-monitored blood glucose values ≤3.0 mmol/L | 12 weeks (total duration of study)
  Number of self-monitored blood glucose values ≤3.0 mmol/L
Severe hypoglycemia | 12 weeks (total duration of study)
  Number of severe hypoglycemic events (defined as severe cognitive impairment requiring external assistance for recovery).
Time spent in hypoglycemia | 8 days (first four and last four days of study)
  Time spent in hypoglycemia (<3.9 mmol/L) assessed by CGM during the first four study days (days without insulin) and the last four study days (days with optimal daily insulin dose).
Time spent in hyperglycemia | 8 days (first four and last four days of study)
  Time spent in hyperglycemia (>10 mmol/L) assessed by CGM during the first four study days (days without insulin) and the last four study days (days with optimal daily insulin dose).
Time spent in normoglycemia | 8 days (first four and last four days of study)
  Time spent in normoglycemia (3.9-10.0 mmol/L) assessed by CGM during the first four study days (days without insulin) and the last four study days (days with optimal daily insulin dose).

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aradottir TB, Bengtsson H, Jensen ML, Poulsen NK, Boiroux D, Jensen LL, Schmidt S, Norgaard K. Feasibility of a New Approach to Initiate Insulin in Type 2 Diabetes. J Diabetes Sci Technol. 2021 Mar;15(2):339-345. doi: 10.1177/1932296819900240. Epub 2020 Jan 15. PMID 31941361